CLINICAL TRIAL: NCT03149211
Title: A Phase III, Randomized, Open-label, Controlled Trial to Investigate the Efficacy and Safety of UB-421 Monotherapy as Substitution for Stable Antiretroviral Therapy in HIV-1 Infected Adults
Brief Title: To Investigate the Efficacy and Safety of UB-421 Monotherapy in HIV-1 Infected Adults
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: project adjustment
Sponsor: United BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UBP-A304-HIV
Record Dates: First submitted 2017-05-02; First posted 2017-05-11 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — UB-421

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): Subjects will receive current standard HAART treatment as the active control group.
  Interventions: Drug: current standard HAART treatment
- Cohort 2 (Experimental): Subjects will receive UB-421 without HAART treatment by intravenous infusion at 25 mg/kg bi-weekly. After 26-week treatment period, subjects will enter 22-week follow-up period with current standard HAART treatment.
  Interventions: Drug: UB-421; Drug: current standard HAART treatment

INTERVENTIONS:
Drug: UB-421 — Subjects will receive 13 doses of the UB-421 by intravenous infusion at 25 mg/kg bi-weekly (Cohort 2, 26 weeks).
  Other Names: dB4C7 mAb
  Arms: Cohort 2
Drug: current standard HAART treatment — Subjects will receive current standard HAART treatment as the active control group.

SUMMARY:
The purpose of this phase III study is to evaluate the efficacy, safety and tolerability of UB-421 monotherapy in suppressing viral rebound in HIV-1 infected adults undergoing antiretroviral treatment interruption.

DETAILED DESCRIPTION:
This is an open-label, Phase III study to evaluate the efficacy, safety and tolerability of UB-421 monotherapy in suppressing viral rebound while replace HAART in virally suppressed HIV-1 infected adults. In this study, approximately 375 subjects on stable HAART treatment will be randomized to receive either continuing HAART treatment alone (Cohort 1) or UB-421 as the monotherapy (Cohort 2) in 1:2 ratio. For Cohort 1, subjects will receive current standard HAART treatment as the active control group. For Cohort 2, UB-421 will be administered to enrolled subjects without HAART treatment in the Cohort 2 during the 26-week treatment period. After treatment period, both cohort 1 and cohort 2 enter 22-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 sero-positive
* Aged 20 years or older
* Were not breastfeeding for women
* Subjects with a negative serum pregnancy test result at screening visit for women of childbearing potential
* Subjects agree on using birth control barrier (female or male condom) during the entire study period
* Subjects sign the informed consent before undergoing any study procedures

Exclusion Criteria:

* Any active infection except for HIV, and required immediate therapy
* Any active AIDS-defining illness per Category B and Category C conditions according to the U.S. Centers for Disease Control and Prevention (CDC) Classification System for HIV Infection
* Any significant diseases (other than HIV-1 infection) or clinically significant findings, including psychiatric and behavioral problems, determined from screening, medical history, and/or physical examination that, in the investigator's opinion, would preclude the subject from participating in this study
* Life expectancy less than 12 months
* Any alcohol or illicit drug used, according to the investigator's opinion, will interfere with the subject's ability to comply with the dosing, visit schedules and protocol evaluations

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants without virologic failure | 24 weeks

SECONDARY OUTCOMES:
Time to virologic failure | 26 weeks
Number of participants with treatment-related adverse events | 48 weeks
Peak concentration of UB-421 in Cohort 2 | 30 weeks
Trough concentration of UB-421 in Cohort 2 | 30 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality, China